CLINICAL TRIAL: NCT00877981
Title: Open Compared to Video-Assisted Minimal-Invasive Parathyroid Surgery in Primary Hyperparathyroidism
Brief Title: Open Versus Video-Assisted Minimal-Invasive Parathyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Lund University (Other); University of Aarhus (Other)
Responsible Party: Ola Hessman, Uppsala University, Dept of Surgical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HPT02
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Primary Hyperparathyroidism
Keywords: hyperparathyroidism; surgery; minimal invasive; videoassited
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hyperparathyroidism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoassited surgery (Active Comparator): In patients randomized to a video-assisted approach, the surgeon has the option to choose either the lateral- (VAPLA) or medial (MIVAP) techniques, both initiated with a 15 mm transverse skin incision. The lateral approach is performed as described by Henry.
  The medial approach is performed using the gasless procedure developed by Miccoli.
  Interventions: Procedure: Minimal invasive Parathyroid surgery
- Open surgery (Active Comparator): Open surgery, a 15 mm transverse skin incision is made close to the site of the parathyroid adenoma indicated by sestamibi scintigraphy.
  Interventions: Procedure: Minimal invasive Parathyroid surgery

INTERVENTIONS:
Procedure: Minimal invasive Parathyroid surgery

SUMMARY:
The aim of the present study was to compare open minimal-invasive parathyroid surgery with video-assisted parathyroidectomy in primary hyperparathyroidism (PHPT) patients with a positive sestamibi scan in a multicentre randomized trial in order to evaluate if videoassisted surgery gave less postoperative pain and if there was a difference in operating time.

DETAILED DESCRIPTION:
The present study is designed to compare open minimal-invasive parathyroid surgery with video-assisted parathyroidectomy in pHPT patients with a positive sestamibi scan in a multicentre prospective randomized trial.

In patients randomized to open surgery, a 15 mm transverse skin incision is made close to the site of the parathyroid adenoma indicated by sestamibi scintigraphy. In case of an enlarged upper parathyroid or dorsally located lower parathyroid, the incision is made anterior to the sternocleidomastoid muscle (SCM) whereas for anterior located lower parathyroids a central incision is chosen.

In patients randomized to a video-assisted approach, the surgeon has the option to choose either the lateral- (VAPLA) or medial (MIVAP) techniques, both initiated with a 15 mm transverse skin incision.

Postoperatively the patients receive a questionnaire for selfdocumentation.Variables recorded include postoperative pain, hypocalcaemic symptoms, breathing problems, cervical discomforts of pressure/globus and voice disturbances. A visual analogue scale (VAS) is used when appropriate. The intake of oral analgesics and calcium medication is also recorded. The questionnaire is used daily for the first four postoperative days, and thereafter weekly for four weeks.

Follow-up is done at 1 and 6 month after surgery, with measurement of plasma calcium and PTH. Continued needs of calcium or vitamin D medication, length of scar, and symptoms or signs of complications are recorded. At the six-month follow-up, patients document their opinion of the cosmetic results and the remaining neck discomfort using a VAS.

Primary outcome measures are postoperative pain and operation time. Secondary outcome measures are complications, persistent or recurrent disease, conversion rates and cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biochemically verified primary hyperparathyroidism and with an unequivocal localisation on sestamibi scintigraphy of a solitary parathyroid adenoma

Exclusion Criteria:

* Negative or equivocal preoperative localization study, familiar HPT, previous neck surgery or neck irradiation, concomitant need of thyroid surgery, pregnancy, suspected ectopic parathyroid localization, or inability to understand information, instructions and/or comply with scheduled follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2003-02; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 4 days
Operating time

SECONDARY OUTCOMES:
complications | 6 months
Persistent or recurrent disease | 6 months
conversion rate
Cosmetic results

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bergenfelz, MD, Ass Prof, Principal Investigator — Department of Surgery, Lund University
Locations (3):
- Unit of Breast and Endocrine Surgery, Surgical Department P, Aarhus University Hospital, Aarhus, Denmark
- Sweden (2):
  - Department of Surgery, Lund University Hospital, Lund
  - Uppsala University Hospital, Dept of surgery, Uppsala

REFERENCES:
- [Derived] Hessman O, Westerdahl J, Al-Suliman N, Christiansen P, Hellman P, Bergenfelz A. Randomized clinical trial comparing open with video-assisted minimally invasive parathyroid surgery for primary hyperparathyroidism. Br J Surg. 2010 Feb;97(2):177-84. doi: 10.1002/bjs.6810. PMID 20035529